CLINICAL TRIAL: NCT05865808
Title: Effects of Sustained Natural Appophyseal Glide Versus Rocababo 6x6 Program in Subjects With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0121
Record Dates: First submitted 2023-05-04; First posted 2023-05-19 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cervicogenic Headache
Keywords: cervical spine; neurological disorder; post-traumatic disorder; secondary headache
MeSH Terms: conditions — Post-Traumatic Headache; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical spine mobilization (Experimental): Subjects in this group will be treated with headache SNAGs
  Interventions: Other: cervical spine mobilization
- Rocabado 6x6 exercises (Active Comparator): Rocabado 6x6 program includes 6 types of exercises which are- rest position of the tongue, TMJ rotation control, upper cervical distraction, axial extension of cervical spine, shoulder girdle retraction, and rhythmic stabilization technique.
  Interventions: Other: Rocabado 6x6

INTERVENTIONS:
Other: cervical spine mobilization — headache SNAGs, 10 repetitions holding for 10 seconds in each glide with a rest time of 30 seconds in between. Eight weeks of treatment session will be provided and assessment of the improvement in cervicogenic headache will done at baseline, after 04, 06 and at the end of 8 week.
  Arms: Cervical spine mobilization
Other: Rocabado 6x6 — The Rocabado 6x6 program includes 6 types of exercises which are- rest position of the tongue, TMJ rotation control, upper cervical distraction, axial extension of cervical spine, shoulder girdle retraction, and rhythmic stabilization technique, which are to be performed 6 times in a day with 6 repetitions of each exercise in each session,
  Arms: Rocabado 6x6 exercises

SUMMARY:
The purpose of this study is to investigate the effects of TMJ directed treatment approach using the Rocabado 6x6 program in patients with cervicogenic headache on the intensity of headache, function of the neck, and quality of life and compare its effectiveness with headache SNAGs which have been proven very effective in treatment of cervicogenic headache.

DETAILED DESCRIPTION:
The efectiveness of Sustained Natural Apophyseal Glide on Flexion Rotation Test, pain intensity, and functionality in subjects with Cervicogenic Headache was evaluated. The research was conducted on five computerized databases PubMed/Medline, Web of Science, PEDro, Lilacs, and Cochrane Library (CENTRAL), using the keywords combination: (sustained natural apophyseal glide OR SNAG OR joint mobilization OR Mulligan) AND (cervicogenic headache) according to PRISMA guidelines. The methodological quality of the included studies was analyzed using the Physiotherapy Evidence Database (PEDro) scale. Eight articles fulflled the eligibility criteria and were included in the review. The selected studies had a methodological quality of 6.6/10 on the PEDro scale and included a total of 357 participants. The SNAG signifcantly improved pain, Flexion Rotation Test and reduced functional symptoms. Conclusion: The available evidence suggests that SNAG may be a relevant intervention for CH.

Effectiveness of different physiotherapy interventions in the management of cervicogenic headache was measured. Spinal mobilization, neural mobilization, and postural correction exercises techniques are physiotherapy interventions used for managing CGH symptoms. 80 participants with diagnosed CGH were recruited and divided into 4 groups. The spinal mobilization group received posteroanterior glide at the spinous and transverse process of C2 and C3 vertebra, lateral glide at affected side of the spinous process of C2 and C3 vertebra and translatoric glide at the transverse process of C1 vertebrae and SNAG. The neural mobilization group received neural mobilization of meninges, brachial plexus, and trigeminal nerve. In postural correction exercises group stretching of tight muscles (rectus capitus posterior, suboccipital, upper trapezeius, scalene, levator scapulae, sternocleidomastoid, pectoralis major/minor muscles) were given. Strengthening and endurance exercises for weak muscles (cervical flexors and deep cervical flexor, rhomboidus, and lower trapezeius muscles) were given. The control group was given normal range of motion exercises for the neck and shoulder region. It was concluded by results that applying any of the three modalities randomly in groups of patients with established CGH resulted in improvements of measured outcomes compared to a control group.

Limited literature is available about TMJ treatment in patients with headaches, and few studies has applied direct interventions to the muscles involved in TMJ movement to relieve headache symptoms. Due to the methodological shortcomings, diversity of interventions and inconsistency of findings, there is currently low certainty that there is an effect of physical therapy for TMJ on concomitant headache intensity compared to control interventions. More studies of higher methodological quality are needed so better conclusions could be taken.Further, till now very few studies have done to prove the effect of Rocabado's approach and neither a single study conducted on its effectiveness for headache.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60 years.
* Unilateral headache that do not shift side with ipsilateral neck pain/stiffness.
* Headache for past 3 months at least once per week.
* Positive flexion rotation test.

Exclusion Criteria:

* Subjects with other type of headache.
* Specific disorders and congenital conditions of cervical spine.
* PT or chiropractic treatment in past 3 months.
* Severe pain, traumatic injury, occlusal splints or any surgery in TMJ area

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 8th week
  Neck Disability Index will be used examine neck pain intensity and cervicogenic headache symptoms.Consists of 10 sections each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.
  Changes from Baseline to 8 weeks.

SECONDARY OUTCOMES:
Headache Impact Test-6 SCALE | 8th week
  The 6-item Headache Impact Test scale will be used to examine headache severity and its adverse effects on social life and functions. Consists of 6 sections that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent Changes from Baseline to 8 weeks.
Flexion Rotation Test | 8th week
  Flexion-Rotation Test to assess rotation range of motion at the level of C1-C2 and confirmed by a cervical range of motion device/goniometer. The reported normal range of rotation during the FRT is 44° to each side and is positive if mobility is restricted by more than 10° or if symptoms occur during the procedure.
  Changes from Baseline to 8 weeks.
Numeric Pain Rating Scale | 8th week
  The numeric pain rating scale for the intensity of pain ranges from 0-10. Zero represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
  Changes from Baseline to 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, phd, Principal Investigator — Riphah International University
Locations (1):
- Zia Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paquin JP, Tousignant-Laflamme Y, Dumas JP. Effects of SNAG mobilization combined with a self-SNAG home-exercise for the treatment of cervicogenic headache: a pilot study. J Man Manip Ther. 2021 Aug;29(4):244-254. doi: 10.1080/10669817.2020.1864960. Epub 2021 Feb 5. PMID 33541242
- [Background] Verma S, Tripathi M, Chandra PS. Cervicogenic Headache: Current Perspectives. Neurol India. 2021 Mar-Apr;69(Supplement):S194-S198. doi: 10.4103/0028-3886.315992. PMID 34003165
- [Background] Cardoso R, Seixas A, Rodrigues S, Moreira-Silva I, Ventura N, Azevedo J, Monsignori F. The effectiveness of Sustained Natural Apophyseal Glide on Flexion Rotation Test, pain intensity, and functionality in subjects with Cervicogenic Headache: A Systematic Review of Randomized Trials. Arch Physiother. 2022 Sep 1;12(1):20. doi: 10.1186/s40945-022-00144-3. PMID 36045409
- [Background] Rani M, Kaur J. Effectiveness of different physiotherapy interventions in the management of cervicogenic headache: a pilot randomized controlled trial. J Man Manip Ther. 2022 Apr;30(2):96-104. doi: 10.1080/10669817.2021.1962687. Epub 2021 Aug 10. PMID 34374330
- [Background] Coskun Benlidayi I MD, Guzel R MD, Tatli U PhD, Salimov F PhD, Keceli O PhD. The relationship between neck pain and cervical alignment in patients with temporomandibular disorders. Cranio. 2020 May;38(3):174-179. doi: 10.1080/08869634.2018.1498181. Epub 2018 Jul 26. PMID 30048225
- [Background] Ghodrati M, Mosallanezhad Z, Shati M, Noroozi M, Moghadam AN, Rostami M, Nourbakhsh MR. Adding Temporomandibular joint treatments to routine physiotherapy for patients with non-specific chronic neck pain: A randomized clinical study. J Bodyw Mov Ther. 2020 Apr;24(2):202-212. doi: 10.1016/j.jbmt.2019.11.004. Epub 2019 Nov 22. PMID 32507146
- [Background] Kang JH. Effects on migraine, neck pain, and head and neck posture, of temporomandibular disorder treatment: Study of a retrospective cohort. Arch Oral Biol. 2020 Jun;114:104718. doi: 10.1016/j.archoralbio.2020.104718. Epub 2020 Apr 18. PMID 32334135
- [Background] Greenbaum T, Dvir Z, Emodi-Perlman A, Reiter S, Rubin P, Winocur E. The association between specific temporomandibular disorders and cervicogenic headache. Musculoskelet Sci Pract. 2021 Apr;52:102321. doi: 10.1016/j.msksp.2021.102321. Epub 2021 Jan 12. PMID 33482538
- [Background] Craciun MD, Geman O, Leuciuc FV, Holubiac IS, Gheorghita D, Filip F. Effectiveness of Physiotherapy in the Treatment of Temporomandibular Joint Dysfunction and the Relationship with Cervical Spine. Biomedicines. 2022 Nov 17;10(11):2962. doi: 10.3390/biomedicines10112962. PMID 36428529
- [Background] Pundkar S, Patil D, Naqvi W. A Comparative Study on Effectiveness of Rocabado Approach and Conventional Physiotherapy on Pain, ROM and QOL in Patients with TMJ Dysfunction. 2021.
- [Background] Corum M. Evaluation of Cervical Dysfunctions in Temporomandibular Disorders. Medical Journal of Bakirkoy. 2021;17(1).
- [Background] La Touche R, Martinez Garcia S, Serrano Garcia B, Proy Acosta A, Adraos Juarez D, Fernandez Perez JJ, Angulo-Diaz-Parreno S, Cuenca-Martinez F, Paris-Alemany A, Suso-Marti L. Effect of Manual Therapy and Therapeutic Exercise Applied to the Cervical Region on Pain and Pressure Pain Sensitivity in Patients with Temporomandibular Disorders: A Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2373-2384. doi: 10.1093/pm/pnaa021. PMID 32181811
- [Derived] Murtza S, Noor R, Bashir MS, Ikram M. Effects of sustained natural apophyseal glides versus rocabado 6 x 6 program in subjects with cervicogenic headache. BMC Musculoskelet Disord. 2024 Feb 22;25(1):169. doi: 10.1186/s12891-024-07290-8. PMID 38389050